CLINICAL TRIAL: NCT03999125
Title: Anti-VEGF Therapy Versus Dexamethasone Implant for Treatment Naive Diabetic Macular Edema: A Randomized Controlled Trial
Brief Title: Anti-VEGF Therapy Versus Dexamethasone Implant for DME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sudhalkar Eye Hospital (Other)
Responsible Party: Principal Investigator, Aditya Sudhalkar, Consultant Vitreoretinal Surgeon, Sudhalkar Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SudhalkarEH
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Clinically Significant Macular Edema Due to Diabetes Mellitus
MeSH Terms: interventions — aflibercept; Ranibizumab; Dexamethasone; Lasers

STUDY DESIGN:
Intervention Model Description: Parallel, multi-arm trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Aflibercept intravitreal injection for CSME
  Interventions: Drug: Aflibercept,
- Group 2 (Other): Ranibizumab Intravitreal Injection for CSME
  Interventions: Drug: Ranibizumab Injection
- Group 3 (Experimental): Dexamethasone Implant for CSME
  Interventions: Drug: Ozurdex Drug Implant Product

INTERVENTIONS:
Drug: Aflibercept, — Primary therapy will be with Aflibercept. If the edema does not respond to the intervention, the patient will be treated with Ranibizumab, Dexamethasone Implant or Laser.
  Other Names: Ranibizumab; Dexamethasone Implant, Laser
  Arms: Group 1
Drug: Ranibizumab Injection — Primary therapy will be with ranibizumab. If the edema does not respond to the intervention, the patient will be treated with Alfibercept, Dexamethasone Implant or Laser.
  Other Names: Dexamethasone Implant, Aflibercept, Laser
  Arms: Group 2
Drug: Ozurdex Drug Implant Product — Primary therapy will be with Ozurdex. If the edema does not respond to the intervention, the patient will be treated with Alfibercept, Ranibizumab or Laser
  Arms: Group 3

SUMMARY:
We look at a randomized comparative study of 2 FDA approved anti-VEGF agents(aflibercept and ranibizumab) and see how they compare against the dexamethasone implant for phakic as well as pseudophakic eyes with treatment naive diabetic macular edema in terms of efficacy and safety over two years.

DETAILED DESCRIPTION:
A randomized, partially masked, observational/interventional trial looking at the efficacy and safety of 2 FDA approved anti-VEGF agents vis-a-vis the dexamethasone implant as primary therapy for treatment naive diabetic macular edema in phakic as well as pseudophakic patients.

Patients with treatment naive clinically significant macular edema will be randomized to receive one of the aforementioned therapies in a 1:1:1 distribution. Primary inclusion criteria are :

Well controlled diabetes(HbA1c<7%) and co-morbidities. Central Subfield Thickness of 300 microns or greater BCVA < or equal to 6/12.

Exclusion Criteria:

Contraindications to the aforementioned drugs Confounding Ocular co-morbidities that can affect visual assessment(except Cataract Grade II or less as per the LOCS III classification) Refusal for enrolment

A comprehensive ocular and systemic examination will be performed along with fundus fluorescein angiography, optical coherence tomography and intraocular pressure measurements with the Goldmann Applanation Tonometer. The BCVA will be recorded using Snellen's chart

Intravitreal injections will be administered using a standardized technique and under strict asepsis. No postoperative antibiotics will be given.

Patients will be followed on postoperative days 1, 7 and then monthly for 2 years.

At each visit, the BCVA, IOP, ocular exam and OCT scans will be performed at each visit.

Patients will be treated as per the guidelines laid out for the treat and extend study. For the dexamethasone implant, re-injections will be allowed first 3 months after the first injection.

Switch therapy is permissible for anti-VEGF agents after 6 months; first to the other anti-VEGF(for 6 more injections) and then to the dexamethasone implant. Rescue Laser therapy is as per physician's description.

Primary outcome measure: The BCVA in each group from baseline to final follow-up at 2 years.

Secondary outcome measure: Change in CST from baseline to years, the number of injections required per group and the complications, if any.

Statistical Analysis will include demographic descriptions, the Shapiro Wilk test to look for normality of distribution, multiple measures ANOVA test, Fisher's exact test, Chi-Square test and paired and unpaired t-test wherever appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Well controlled diabetes(HbA1c<7%) and co-morbidities. Central Subfield Thickness of 300 microns or greater BCVA < or equal to 6/12.

Exclusion Criteria:

* Contraindications to the aforementioned drugs Confounding Ocular co-morbidities that can affect visual assessment(except Cataract Grade II or less as per the LOCS III classification) Macular ischemia or proliferative Disease Refusal for enrolment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-25 (Estimated); Primary Completion 2021-06-24 (Estimated); Study Completion 2023-06-24 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 2 years
  BCVA measured at baseline and final follow-up

SECONDARY OUTCOMES:
Central Subfield Thickness | 2 years
  Change in CST over 2 years
Complications | 2 years
  Complications in each group
Injection Count | 2 years
  Number of injections in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Alphavision Augenzentrum, Bremerhaven, City state Bremen, Germany

IPD SHARING:
Plan to Share IPD: Yes
All details of FFA, OCT, BCVA and IOP
Supporting Information: Study Protocol, SAP
Time Frame: Upon completion of study
Access Criteria: Will be provided only to Ophthalmologists